CLINICAL TRIAL: NCT07327502
Title: Cefazolin Distribution in Mediastinum After Heart Surgery in Children Using a Microdialysis Probe.
Brief Title: Antibiotics Distribution Study in Peripheral Compartments: Contribution of Microdialysis
Acronym: Antimidis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP241591; 2025-521988-13 (EudraCT Number)
Record Dates: First submitted 2025-12-08; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Children in Cardiac Intensive Care Requiring Surgery for Congenital Heart Disease
Keywords: Cefazolin; Cardiac surgery; Mediastinitis; Microdialysis
MeSH Terms: conditions — Mediastinitis | interventions — Microdialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cefazolin measurements (Experimental): Microdialysis probe placement and blood drawings to measure cefazolin concentration in mediastinum tissue and in plasma.
  Interventions: Procedure: Microdialysis probe placement; Procedure: Microdialysis and Plasma samples

INTERVENTIONS:
Procedure: Microdialysis probe placement — Microdialysis probe is placed at the end of cardiac surgery in mediastinum and used during 36 hours for tissue samples until withdrawal.
Procedure: Microdialysis and Plasma samples — 26 Cefazolin Free tissue concentrations 6 total plasma concentrations

SUMMARY:
Postoperative mediastinitis is an important cause of postoperative morbidity in children. The main objective of this study is to describe the distribution of cefazolin, using as surgical antibiotic prophylaxis, in the mediastinal compartment in children after cardiac surgery for congenital heart disease. The investigators aims to build a population pharmacokinetic model of cefazolin using plasma and tissue concentrations in order to optimize and individualize cefazolin dosing regimens. Cefazolin tissue pharmacokinetics will use a microdialysis procedure.

DETAILED DESCRIPTION:
Children with congenital heart disease are very fragile during the postoperative period and at risk of life-threatening mediastinitis due to various factors: post-extracorporeal circulation inflammation, frequent organ failure, possible delayed thorax closure. These patients are at risk of unpredictable pharmacokinetics alteration and inter-individual variability of the drug tissue: significant fluid intake, drug metabolism and elimination functions alteration, extracorporeal circulation. The effective prevention of postoperative mediastinitis in this population is therefore a major issue and challenge. Studying the distribution of cefazolin in the mediastinum and identifying the factors of inter-individual variability would improve the prevention of this pathology by optimizing the dosing.

During cardiac surgery, a microdialysis probe is placed by the surgeon in the mediastinum. The outgoing fluid will be collected every 30 minutes to every 2 hours, for approximately 28 hours. Six plasma samples will be drawn over these 28 hours to measure plasma concentrations. The probe's recovery will then be calculated and the probe will be removed up to 36 hours after insertion.

ELIGIBILITY:
Inclusion Criteria:

* Child aged over 6 months and under 6 years
* Hospitalized in pediatric cardiac intensive care after cardiac surgery for congenital heart disease.
* Selected congenital heart diseases: ventricular septal defect auricular septal defect, pulmonary stenosis, tetralogy of Fallot
* Surgery with median sternotomy and intraoperative cardiopulmonary bypass
* Intraoperative antibiotic prophylaxis with cefazolin
* Patient affiliated with a social security plan or eligible
* whose two parents or legal guardians have accepted and signed the study consent

Exclusion Criteria:

* Emergency cardiac surgery
* Patient already enrolled in the study
* Patient who has previously undergone cardiac surgery
* Patient with haemostasis disorders or immune deficiency
* Patient with bacterial colonization indicating antibiotic prophylaxis other than cefazolin
* Participation in another interventional research study

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Total clearance | 36 hours
  Pharmacokinetics of cefazolin total clearance in children after cardiac surgery and inter-individual variability.
Distribution volume | 36 hours
  Pharmacokinetics of cefazolin distribution volume in children after cardiac surgery and inter-individual variability.
Inter-compartmental clearance | 36 hours
  Pharmacokinetics of cefazolin inter-compartmental clearance in children after cardiac surgery and inter-individual variability.

SECONDARY OUTCOMES:
Monte Carlo simulations and dosing optimization | 36 hours
  Monte Carlo simulations performed using the model with SimulX (version 2024R1) and R (version 4.4.2) softwares. Probability of attainment of PK/PD target (100 % ƒT > 4xCMI) with simulated dosing regimens No patient data is required for this step.
post-operative mediastinitis occurrence | Month 1
  Assess the relationship between tissue exposure and clinical outcome: occurrence of post-operative mediastinitis

CONTACTS AND LOCATIONS:
Overall Officials: Margaux Pontailler, MD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants Malades, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Himebauch AS, Sankar WN, Flynn JM, Sisko MT, Moorthy GS, Gerber JS, Zuppa AF, Fox E, Dormans JP, Kilbaugh TJ. Skeletal muscle and plasma concentrations of cefazolin during complex paediatric spinal surgery. Br J Anaesth. 2016 Jul;117(1):87-94. doi: 10.1093/bja/aew032. PMID 27317707
- [Background] Andreas M, Zeitlinger M, Wisser W, Jaeger W, Maier-Salamon A, Thalhammer F, Kocher A, Hiesmayr JM, Laufer G, Hutschala D. Cefazolin and linezolid penetration into sternal cancellous bone during coronary artery bypass grafting. Eur J Cardiothorac Surg. 2015 Nov;48(5):758-64. doi: 10.1093/ejcts/ezu491. Epub 2014 Dec 18. PMID 25527166